CLINICAL TRIAL: NCT02095535
Title: The Minimum ChloraPrep Drying Time Before Neuraxial Anesthesia in Elective Cesarean Delivery Patients - Prospective Observational Study
Brief Title: Chlorhexidine Drying Time
Acronym: Chlorhexidine
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Vit Gunka, Principle Investigator, University of British Columbia
Other Study IDs: H14-00623
Record Dates: First submitted 2014-03-19; First posted 2014-03-24 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-04

CONDITIONS: Drying Time
Keywords: obstetric patients; chloraprep; chlorhexidine; drying time
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: All study participants
  Interventions: Drug: Chlorhexidine gluconate

INTERVENTIONS:
Drug: Chlorhexidine gluconate — antiseptic
  Other Names: Chloraprep

SUMMARY:
Before a patient gets a spinal/epidural, their lower back is cleaned with an antiseptic solution diluted in alcohol called ChloraPrep. ChloraPrep must completely dry before starting the anesthetic procedure. It is not known how much time is needed for the solution to completely dry. The investigators aim to determine this.

As the ChloraPrep dries, the alcohol is converted into vapour. The investigators will be using a PPBRae 3000 device to detect small amounts of vapours in the air. As the ChloraPrep dries it gives off less and less vapour. The investigators will use this diminishing vapour concentration to determine when drying is complete.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* At full term
* Due to have a cesarean section under spinal or epidural anesthesia
* 19 to 40 years of age

Exclusion Criteria:

* Allergy to certain antiseptic solutions
* Not suitable for a spinal/epidural anesthetic
* Have a significant amount of hair on lower back

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Elective cesarean patients at BC Women's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vit Gunka, MD FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Period: Recruitment
Arm/Group | Study Group
Started | 20
Completed | 18
Not Completed | 2
Not completed — Protocol Violation | 2
Period: Analysis
Arm/Group | Study Group
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 18

OUTCOME MEASURES:

1. Primary Outcome: Length of Drying Time
Description: Length of drying time from when Chloraprep solution is applied to skin to when skin is deemed dry.
Time Frame: At Chloraprep application
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Study Group
Number analyzed (Participants) | 18
seconds | 123 (32)

ADVERSE EVENTS:
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
* Small sample size
* Severe methodological assumptions (i.e. measuring of ChloraPrep drying time, lack of gold standard to assess wetness/dryness
* Patient's variables could influence wetness
* No enrollment of high BMI patients with skin folds

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No